CLINICAL TRIAL: NCT01416519
Title: Incentive Spirometry Decreases Respiratory Complications After Myocardial Revascularization
Brief Title: Physiotherapy Technique Decreases Respiratory Complications After Cardiac Operation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santa Casa de Votuporanga (Other)
Responsible Party: Principal Investigator, Marcos Aurelio Barboza de Oliveira, M.D., Santa Casa de Votuporanga
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U1111-1123-6476; 0035/2010 (Other: Ethics committee)
Record Dates: First submitted 2011-08-12; First posted 2011-08-15 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Pneumonia; Pleural Effusion; Atelectasis
Keywords: Continuous Positive Airway Pressure; Cough; Oxygen Inhalation Therapy
MeSH Terms: conditions — Pneumonia; Pleural Effusion; Pulmonary Atelectasis; Cough | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): After extubation, starting non-invasive ventilation with face mask (1 hour) followed by assisted cough maneuver. Total of 18 calls in 72 hours distributed as long the patient was extubated.
  Interventions: Procedure: Continuous Positive Airway Pressure (CPAP) facial mask
- Group 2 (Experimental): After extubation, starting early supplemental oxygen with Venturi (FiO2 50%) with gradual weaning, applying assisted deep inspiration technique with Voldyne(R) with four sets of 10 repetitions and assisted cough maneuver. Total of 18 calls in 72 hours distributed as long the patient was extubated.
  Interventions: Procedure: Assisted deep inspiration technique

INTERVENTIONS:
Procedure: Continuous Positive Airway Pressure (CPAP) facial mask — After extubation, starting non-invasive ventilation with face mask (1 hour) followed by assisted cough maneuver. Total of 18 calls in 72 hours distributed as long the patient was extubated.
  Other Names: CPAP
  Arms: Group 1
Procedure: Assisted deep inspiration technique — After extubation, starting early supplemental oxygen with Venturi (FiO2 50%) with gradual weaning, applying assisted deep inspiration technique with Voldyne(R) with four sets of 10 repetitions and assisted cough maneuver. Total of 18 calls in 72 hours distributed as long the patient was extubated.
  Other Names: Voldyne
  Arms: Group 2

SUMMARY:
The objective of this study is to assess whether there is a difference between a care protocol with the use of incentive spirometry (Voldyne ®) and another with the application of NIV (non invasive ventilation with single-level pressure) as a form of therapy. The main focus of the study is to determine the incidence of pulmonary complications in each technique.

DETAILED DESCRIPTION:
Coronary artery bypass graft (CABG) can prolong and improve the quality of life of patients with ischemic coronary syndrome but with the advancement of medical intervention to eligible patients for this procedure are those with more comorbidities where conservation and palliative therapies have been tried without success.

Patients undergoing CABG often develop pulmonary complications such as atelectasis, restrictive ventilatory defect, decreased lung compliance, increased shunt and changes in gas exchange leading to probable hypoxemia. In an attempt to reduce the harmful effects and pulmonary complications arising from surgical procedures is instituted extensive physiotherapy program that tracks and monitors such patients from the preoperative to the postoperative immediate transfer to the ward and hospital discharge.

The objective of this study is to assess whether there is a difference between a care protocol with the use of incentive spirometry (Voldyne ®) and another with the application of NIV (non invasive ventilation with single-level pressure) as a form of therapy. The main focus of the study is to determine the incidence of pulmonary complications in each technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for elective coronary artery bypass surgery who agreed to participate and signed the informed consent.

Exclusion Criteria:

* patients with hemodynamic instability during the physiotherapy care
* those who fail to complete all visits to the proposed protocol (whatever the reason)
* extubation after 12 hours of ICU admission
* major intraoperative hemorrhage
* major bleeding in ICU requiring return to the operating room
* cardiopulmonary arrest
* contraindication to positive pressure (undrained pneumothorax, bronchopleural fistula, hemoptysis, vomiting) or intolerance to the method

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary complications | 72 hours
  Occurrence of pulmonary complications such as pneumonia, atelectasis or pleural effusion diagnosed with chest X-rays by ICU doctor.

SECONDARY OUTCOMES:
Exams | 72 hours
  Assessment of (Sat O2) capillary saturation, (ABG) arterial blood gases.

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Aurelio Barboza de Oliveira, MD, Principal Investigator — Santa Casa Votuporanga
Locations (1):
- Santa Casa Votuporanga, Votuporanga, São Paulo, Brazil